CLINICAL TRIAL: NCT02396563
Title: Effect of Epidural Analgesia on the Length of Labor and Delivery and Fetal Outcomes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Cagliari (Other)
Responsible Party: Principal Investigator, Stefano Angioni, Associate Professor, University of Cagliari
Other Study IDs: LABORCA
Record Dates: First submitted 2015-03-11; First posted 2015-03-24 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Labor; Epidural Analgesia; Nulliparous
MeSH Terms: interventions — Analgesia, Epidural; Ropivacaine

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- epidural analgesia: women in labor with epidural analgesia
  Interventions: Procedure: epidural analgesia; Drug: Ropivacaine
- no epidural analgesia

INTERVENTIONS:
Procedure: epidural analgesia
  Groups: epidural analgesia
Drug: Ropivacaine
  Groups: epidural analgesia

SUMMARY:
The purpose of this study is to determine if there is a difference in the duration of the first and second stage of labor in nulliparous women , with or without epidural analgesia. The investigators hypothesize that the duration of the first stage of labor will be no different in nulliparous patients, while the duration of the second stage will be longer in patient with analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous
* > 18 years old
* term (>37 weeks gestation)
* singleton
* vertex pregnancies

Exclusion Criteria:

* Non-vertex presentation
* cervical dilation > 4.0cm

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women who come to the Gynecological nd obstetric Department of University Hospital to deliver
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
duration of labor | Onset of contractions or rupture of membrances to delivery

SECONDARY OUTCOMES:
Presence or absence of fetal heart rate decelerations | Time of first analgesic dose to 60 minutes
fetal tachycardia | Time of first analgesic dose to 60 minutes